CLINICAL TRIAL: NCT06657872
Title: Local Anesthesia With Schelin Catheter in Rezum Treatment: a Randomized Controlled Trial
Acronym: LOCALVAPOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCAPHM24_0263; 2024-A01800-47 (Other: ANSM)
Record Dates: First submitted 2024-10-21; First posted 2024-10-26 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: REZUM; MIST; general anesthesia; local anesthesia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- general anesthesia (Active Comparator): REZUM procedure under general anesthesia
  Interventions: Procedure: water vapor therapy under general anesthesia
- Local anesthesia (Active Comparator): REZUM procedure under local anesthesia
  Interventions: Procedure: water vapor therapy under local anesthesia

INTERVENTIONS:
Procedure: water vapor therapy under general anesthesia — Water vapor procedure will be performe under conscious intravenous sedation with anesthesia team
  Arms: general anesthesia
Procedure: water vapor therapy under local anesthesia — Water vapor procedure will be performe under local anethesia administrated with Schelin® catheter via the trans-urethral route : injection of 20cc of lidocaine 2% intra-prostatically via the schelin catheter at 4 injection points (3cc at 1h, 3cc at 11h, 7cc at 4h, and 7cc at 8h).
  Arms: Local anesthesia

SUMMARY:
In a pilot study, water vapor therapy (RezumTM, Boston Scientific Corporation, Marlborough, MA) was proposed as a minimally invasive procedure for benign prostatic hyperplasia, but often requiring oral ± intravenous sedation or a transrectal prostatic block. Therefore, pain management during Rezum therapy remains a challenge and may lead to the use of pain control protocols and general anesthesia, limiting in some ways the concept of a minimally invasive ambulatory surgical approach. The Schelin® catheter (ProstaLund AB, Lund, Sweden), approved by the European Medicines Agency, is a device for injecting analgesic drugs directly into the prostate via the trans-urethral route, providing more effective local anesthesia and avoiding the need for transrectal route or general anesthesia. This catheter is therefore of crucial importance in offering to our patients an ultra-minimally invasive treatment, associated with a reduction in room occupancy time, outpatient surgery time, a procedure performed independently of the anesthesia team, and for the patient, an accelerated post-operative recovery. Our hypothesis is that the REZUM procedure under local anesthesia could be associated with a >20% reduction in operating room occupancy time compared to procedures performed under general anesthesia.

DETAILED DESCRIPTION:
Benign prostatic hyperplasia (BPH) is a common age-related pathology, affecting almost one in three men over the age of 50. It is responsible for voiding disorders in men, which can significantly impair quality of life. Briefly, drug treatment is currently used as first-line therapy; in the event of primary or secondary failure, surgery may be indicated. Over the past 25 years, a number of minimally invasive surgical therapies (MIST) have been developed for the treatment of male voiding disorders associated with BPH. MIST should enable rapid and lasting improvement in symptoms and quality of life, preservation of sexual function in contrast to conventional surgical techniques, rapid return to normal daily activity, and a minimal side-effect profile, thus enabling outpatient management. One of the many advantages of these techniques is to avoid the need for general anaesthesia, both for the growing cohort of elderly patients and for younger patients wishing to return to work quickly. In its pilot study, water vapor thermal therapy (RezumTM, Boston Scientific Corporation, Marlborough, MA) was proposed as a minimally invasive procedure, but often requiring oral ± intravenous sedation or a transrectal prostatic block. Therefore, pain management during Rezum therapy remains a challenge and may lead to the use of pain control protocols and general anesthesia, in some ways limiting the concept of a minimally invasive ambulatory surgery approach. In addition, the use of general anesthesia requires the presence of a dedicated anesthesia team, and adds to the burden of the patient journey (pre-operative anesthesia consultation, exposure to anesthetic drugs, passage to recovery room, slower post-operative recovery). From a surgical point of view, recourse to general anesthesia during Rezum treatment adds to an already saturated operative schedule, with significantly increased room occupancy time, for a Rezum therapy whose average operating time is 5 minutes. The Schelin® catheter (ProstaLund AB, Lund, Sweden), approved by the European Medicines Agency, is a device for injecting analgesic drugs directly into the prostate via the transurethral route, providing more effective local anesthesia and avoiding the need for transrectal or general anesthesia. This catheter is therefore of crucial use in offering our patients an ultra-minimally invasive treatment, which can be associated with a reduction in room occupancy time, time spent in outpatient surgery, a procedure performed independently of the anesthesia team, and for the patient, an accelerated post-operative recovery.

By delivering the Rezum treatment via the Schelin catheter, our hypothesis is a significant reduction (>20%) in room occupancy time in the operating room, associated with accelerated post-operative recovery for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for symptomatic benign prostatic hyperplasia (BPH)
* Men between 45 and 80 years of age
* IPSS > 13
* Qmax <15 ml/s
* Prostate volume between 30 and 80 g on ultrasound
* Patient able to understand study details, benefits and risks
* Patient able to give informed consent
* Beneficiary of or affiliated to the French social security system
* Patient having signed an informed consent form

Exclusion Criteria:

* Patients with a history of prostate cancer
* Patient with history of BPH surgery
* Patients with a history of neurological bladder disease
* Patient with history of urethral stricture
* Patient with history of penile implants
* Patient with history of pelvic irradiation
* Patient with a symptomatic urinary tract infection in the 10 days prior to surgery
* Presence of bladder stones on ultrasonography
* Patient allergic to lidocaine 2% or any medication used in the pre-operative protocol (anxiolytics, analgesics and non-steroidal anti-inflammatory drugs)
* Patient under guardianship or curatorship
* Protected patient, deprived of liberty
* Patient with a neurological and/or psychiatric disorder making it impossible to understand the terms of the study and to sign an informed consent form

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study focus on benign prostatic hyperplasia
Enrollment: 24 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2026-11-24 (Estimated); Study Completion 2026-11-24 (Estimated)

PRIMARY OUTCOMES:
Comparison of the operating room occupancy time between the 2 groups | Visit 2: surgery
  Operating room occupancy time during REZUM procedure

SECONDARY OUTCOMES:
Comparison of the quality of recovery after surgery between the 2 groups | 24h after surgery
  Quality of recovery-15 scores (QoR-15)
Comparison of the pain post-surgery between the 2 groups | 1 hour, 2 hours and 24 hours after surgery
  Numerical pain rating scale (0-10)
Success rate of the local anesthesia for the REZUM procedure | intraoperative
  * Number of patients with intraoperative anesthesia changes
  * Numerical pain rating scale (0-10) during surgery
Comparison of functional results between the 2 groups | 3 months post-surgery
  urinary function assessment:
  * International Prostate Symptom Score
  * International Prostate Symptom Score - Quality of Life
  * Uriflometry (Qmax)
  Sexual function assessment:
  * International Index of Erectile Function
  * Male Sexual Health Questionnaire
Comparison of the average number of side-effects post-surgery between the 2 groups | 30 days post-surgery
  Post-operative side effects reported using the Clavien-Dindo classification

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'urologie, Hôpital Nord (AP-HM), Marseille, France

IPD SHARING:
Plan to Share IPD: No